CLINICAL TRIAL: NCT05572437
Title: Perioperative Effect of Music in Patients Undergoing General Anesthesia
Acronym: EMBAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra, Principal Investigator, Dr. Negrin University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-370-1
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Perioperative Anxiety; Postoperative Pain
Keywords: Anxiety, Perioperative, Insomnia
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The randomization of the patients will be carried out by a collaborating researcher through a computer program (Excel 2016) at the time of inclusion in the study. This collaborating researcher will not be able to be present at the surgical intervention and will contact the nursing staff by telephone, indicating which patient should be given music therapy upon arrival in the pre-surgery room.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: El investigador responsable de la recogida de los datos a partir del informe clínico de los anestesiólogos responsables del manejo clínico intra y postoperatorio de los pacientes no sabrá qué pacientes han sido incluidos en el grupo Intervención.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients randomized to the control group will be assessed for preoperative anxiety using the APAIS scale in the preoperative room and assessment of insomnia using the ISI scale both in the PACU and on the 1st day in the hospital ward. Pain assessment will be measured using the VAS scale in the PACU and on the first day on the hospital ward.
- Intervention Group (Experimental): Patients randomized to the treatment with music group (classical music), after assessment of anxiety using the APAIS scale, will be given headphones and classical music will be played from their stay in the pre-surgery room, during surgery and in the PACU.
  Interventions: Device: Music Therapy

INTERVENTIONS:
Device: Music Therapy — Patients randomized to the treatment with music group (classical music), after assessment of anxiety using the APAIS scale, will be given headphones and classical music will be played from their stay in the pre-anesthesia room, during surgery and in the PACU.
  Arms: Intervention Group

SUMMARY:
Anxiety is a transient emotional state characterized by feelings of tension, apprehension, nervousness, fear, and heightened activation of the autonomic nervous system in response to a specific current or potential event or situation. Music therapy is a cost-effective and safe intervention applied to health care, that has been incorporated into different branches of medicine, including anesthesiology, showing economic benefits and as an adjunct to pharmacological therapy, allowing the use of lower doses of perioperative drugs, thus reducing their deleterious effects. The main objective of this randomized clinical trial is to evaluate whether the application of music during the perioperative period reduces perioperative anxiety in patients undergoing general and digestive surgery under general anesthesia.Patients between 18 and 60 years of age, classified according to the American Society of Anesthesiologists (ASA) I-IV, scheduled for general surgery and who have signed the informed consent, will be randomized to receive music therapy in the immediate perioperative period or not. Perioperative anxiety, stay in the PACU, incidence of postoperative pain and intraoperative opioid consumption will be compared between both groups.

DETAILED DESCRIPTION:
Anxiety is a transient emotional state characterized by feelings of tension, apprehension, nervousness, fear, and heightened activation of the autonomic nervous system in response to a specific current or potential event or situation. Music therapy is a cost-effective, non-invasive and safe intervention applied to health care, whose boom has grown gradually in recent years until it has been incorporated into different branches of medicine, including anesthesiology , showing economic benefits and as an adjunct to pharmacological therapy, since it allows the use of lower doses of some drugs, thus reducing their deleterious effects. The main objective of this randomized clinical trial is to evaluate whether the application of music during the perioperative period reduces perioperative anxiety in patients undergoing general and digestive surgery under general anesthesia. Patients between 18 and 60 years of age, classified according to the American Society of Anesthesiologists (ASA) I-IV, scheduled for general surgery and who have signed the informed consent, will be randomized to receive music therapy in the immediate perioperative period or not. Patients randomized to the control group will be assessed for preoperative anxiety using the APAIS and the STAI scales in the preoperative room and assessment of insomnia using the ISI scale both in the PACU and on the 1st day in the hospital ward. Pain assessment will be measured using the VAS scale in the PACU and on the first day in the hospital ward. Patients randomized to the treatment with music group (classical music), after assessment of anxiety using the APAIS and STAI scales, will be given headphones and classical music will be played from their stay in the pre-surgery room, during surgery and in the PACU.All patients will have their anxiety assessed in the pre-anesthesia room and insomnia assessed both in the PACU and on the 1st day in the hospital ward. Pain assessment will be measured in the PACU and on the first day in the hospitalization ward. Perioperative anxiety, stay in the PACU, incidence of postoperative pain and intraoperative opioid consumption will be compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age and under 60 years of age
* Classification of the American Society of Anesthesiologists (ASA) I-IV
* Intervened on a scheduled basis for general surgery.
* Signed informed consent prior to surgery.

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Patients under 18 years of age or incapable of giving their consent.
* ASA V.
* History of hypersensitivity to contact devices
* Patients with total hearing impairment
* Patients with substance abuse use disorders
* Patients with cognitive deficit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Perioperative anxiety | from the arrival to the preanesthesia room to the 4 postoperative hour
  Specific anxiety questionnaires (APAIS, STAI) will be applied on arrival at the pre-anesthesia room, prior to anesthetic induction and after arrival at the post-anesthetic recovery unit.

SECONDARY OUTCOMES:
Postoperative pain | From the first postoperative hour to the 4th postoperative hour.
  Postoperative pain will be assessed using the visual analog scale in the immediate postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Becerra, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Doctor Negrín
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No
IPD are to be shared with other researchers when required once the study is completed and global data are published.